CLINICAL TRIAL: NCT05415631
Title: Augmented Bladder Tumor Detection Using the Bladder-Portable Artifact Detection System: A Multicentric Prospective Analytic Study Using Real Time Based Artificial Intelligence (IA).
Brief Title: Augmented Bladder Tumor Detection Using Real Time Based Artificial Intelligence
Acronym: Bladder-PAD
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2022_843_0014
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-05

CONDITIONS: Bladder Cancer; Cystoscopy; Artificial Intelligence
Keywords: Bladder Cancer; cystoscopy; Artificial Intelligence
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today the standard for the diagnosis and monitoring of bladder tumors is bladder endoscopy. The performance of this exam is not perfect. With this work, based on artificial intelligence, the investigators wish to combine endoscopy with a complementary diagnostic tool in order to improve patient care. The main objective will be to reduce diagnostic errors / wanderings in patients treated or followed for bladder tumors, by imposing a new standard of diagnostic bladder mapping (high PPV and VPN, high precision)(primary purpose diagnostic). The secondary objective will be to homogenize and systematize the descriptive part of the lesions, and to use AI to better characterize tumor aggressiveness. The final objective being to validate a new precision tool (diagnostic companion) essential for developing and standardizing the therapeutic management of bladder tumors (correcting inter-observer heterogeneity).

In this project, video frame will be first extracted from our dataset of cystoscopy videos hosted in in the Next Cloud Recherche. Selected medical image will be segmented and analyzed using our pre-trained CNN model with a feature detection algorithm to obtain features.

Data will be analyzed on both patient and lesion levels. The study will assess the Bladder-PAD accuracy on the detection of bladder tumors, and its ability to predict tumor risk of recurrence and progression.

ELIGIBILITY:
Inclusion Criteria:

* unifocal primary or recurrent suspected bladder cancer with tumor size less or equal than 3 cm
* multifocal primary or recurrent suspected bladder cancer less or equal than 5 lesions and with tumor size less or equal than 3 cm.

Exclusion Criteria:

* Evidence of more than 5 tumors or more than 3 cm
* computed tomography/cystoscopy suspect of muscle-invasive bladder cancer (cT2 or higher)
* computed tomography/magnetic resonance evidence of distant metastases (lymphatic or organic)
* Exclusion criteria will include gross hematuria and bacillus Calmette-Guerin (BCG) treatment or chemotherapy within 3 months of inclusion
* An exception will be made if patients had received only a single course of chemotherapy immediately following TUR
* Patients objecting to the use of their data in the context of research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated for bladder cancer, and prospectively collected at the time of cancer diagnosis, from 01 February 2022 to 01 February 2027
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Tumor detection rate of white light cystoscopy | one day
Tumor detection rate of Bladder-PAD cystoscopy | one day
Tumor false detection rate of white light cystoscopy | one day
Tumor false detection rate of Bladder-PAD cystoscopy | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No